CLINICAL TRIAL: NCT00534690
Title: Lowering VT and Increasing PEP During One-Lung Ventilation (OLV), Impact on Oxygenation
Brief Title: Does PEP Compensate the Reduction of Tidal Volume During One Lung Ventilation?
Acronym: REVOLU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Julie Boussuge, University Hospital, Bordeaux
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHUBX 2007/06
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2010-01

CONDITIONS: Lung Neoplasms; Pulmonary Disease
Keywords: Pulmonary disease; Intubation, Intratracheal; Positive-pressure ventilation
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases | interventions — One-Lung Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other)
  Interventions: Procedure: One-Lung ventilation
- 2 (Other)
  Interventions: Procedure: One-Llung ventilation

INTERVENTIONS:
Procedure: One-Lung ventilation — Low Vt, High PEP
  Arms: 1
Procedure: One-Llung ventilation — High Vt, low PEP
  Arms: 2

SUMMARY:
During general anesthesia, airway closure and the formation of atelectasis impair oxygenation. During one-lung ventilation, large tidal volumes are used to resume atelectasis with a risk of regional over distension and Ventilator-Induced Lung Injury (VILI). The reduction in TV should reduce the occurrence of VILI but lead to a consistent alveolar derecruitment. This harmful effect may be counteracted by PEP. We, therefore, study the impact on oxygenation, of increasing PEP during OLV, in order to maintain alveolar recruitment when TV is reduced.

DETAILED DESCRIPTION:
Approval Status: Approved Approval Number: 2007-06 Board Name: CPP Sud Ouest et Outre-Mer 3 Board Affiliation: French Ministry of Health (DGS) Phone: Email: cpp.soom3@orange.fr No France: Afssaps - French Health Products Safety Agency

During general anesthesia, airway closure and the formation of atelectasis impair oxygenation. During one-lung ventilation, large tidal volumes are used to resume atelectasis with a risk of regional over distension and Ventilator-Induced Lung Injury (VILI). The reduction in TV should reduce the occurrence of VILI but lead to a consistent alveolar derecruitment. This harmful effect may be counteracted by PEP. We, therefore, study the impact on oxygenation, of increasing PEP during OLV, in order to maintain alveolar recruitment when TV is reduced.

A recent study reported that mechanical ventilation with large intraoperative TV is associated with an increased risk of post-pneumonectomy respiratory failure. Indeed, large TV during OLV may lead to Ventilator-Induced Lung Injury (VILI) with the creation of alveolar stretch injury and the development of permeability pulmonary edema. The reduction in TV should reduce the occurrence of VILI but lead to a consistent alveolar derecruitment. This harmful effect may be counteracted by PEP. Therefore, once TV is reduced, PEP may play a key role in minimizing lung collapse and preventing lung units from repeated opening and collapse phases. Such "protective" ventilatory strategy may be proposed if it does not lead to hypoxemia during exclusion. We, therefore, study the impact on oxygenation, of increasing PEP in order to maintain recruitment, keeping Pplat constant when TV is reduced. We will compare, in each patient without severe pulmonary obstructive disease (FEV1 and FEV1 /CV > 70%), two strategies of ventilation with two different levels of TV and PEP, but keeping the same Pplat :

After induction of anesthesia, fiberoptic bronchoscopy confirms the correct position of the tube. Anesthesia is maintained with sevoflurane with a BIS® objective between 45 and 55. Boluses of sufentanyl and cisatracurium are done when clinically necessary. Patients are ventilated in VCV with a ZEUS® respiratory device (Dragger, Germany). Before incision, patients are switched to one-lung ventilation in the lateral position. The tidal volume (TV) is 8 ml/kg of ideal body weight, with a maximal plateau pressure limited to 32 cm H2O. The ventilatory frequency is adjusted in order to maintain end tidal concentrations of carbon dioxide (PetCO2) between 30 to 35 mmHg. 5 cmH2O of positive end expiratory pressure (PEP) is used, and the inspired oxygen fraction is adjusted in order to maintain the pulse oxymetry above 95%. During OLV, if SpO2 decreases to less than 90% with 100% of inspired oxygen fraction, surgery is temporarily stopped to resume two lungs ventilation until SpO2 recover at least 95%. If necessary, a continuous positive airway pressure (CPAP) with 5 cm H2O of oxygen is maintained to provide the non dependent lung. Datas are recorded when the chest is opened. The alveolar pressures and the inspiratory and expiratory flow time curves are monitored. After a period of 15 min, the two strategies are compared in a random order :

* TV of 8 ml/kg of ideal body weight and a PEP of 5 cmH2O during 10 minutes
* TV of 5 ml/kg and a PEP level in order to keep the same plateau pressure during 10 minutes.

Arterial blood gases are measured after 10 minutes using each strategy and before any vessels are ligated. The occurrence of PEPi is detected on the expiratory flow time curve.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Open-chest thoracotomy for pulmonary resection
* oral consent

Exclusion Criteria:

* Severe obstructive disease (FEV1 or FEV1 /CV < 70%)
* Patient who don't tolerate a one-lung ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2007-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
PaO2/FiO2 after 10 minutes of each strategy | 15 minutes after selective intubation and 10 minutes after the beginning of each ventilation type.

SECONDARY OUTCOMES:
Occurrence of intrinsic PEP. | Peroperative period
Haemodynamic side effects: decrease of more than 20% of the arterial systolic blood pressure | peroperative period

CONTACTS AND LOCATIONS:
Overall Officials: Hadrien ROZE, Dr, Principal Investigator — University Hospital, Bordeaux; Paul PEREZ, Dr, Study Chair — University Hospital (USMR), Bordeaux
Locations (1):
- Département d'Anesthésie-Réanimation II, Groupe Hospitalier Sud, CHU de Bordeaux, Pessac, France

REFERENCES:
- [Background] Fernandez-Perez ER, Keegan MT, Brown DR, Hubmayr RD, Gajic O. Intraoperative tidal volume as a risk factor for respiratory failure after pneumonectomy. Anesthesiology. 2006 Jul;105(1):14-8. doi: 10.1097/00000542-200607000-00007. PMID 16809989
- [Background] Gothard J. Lung injury after thoracic surgery and one-lung ventilation. Curr Opin Anaesthesiol. 2006 Feb;19(1):5-10. doi: 10.1097/01.aco.0000192783.40021.c1. PMID 16547427
- [Background] Slinger P. Pro: low tidal volume is indicated during one-lung ventilation. Anesth Analg. 2006 Aug;103(2):268-70. doi: 10.1213/01.ane.0000223701.24874.c8. No abstract available. PMID 16861400
- [Background] Senturk M. New concepts of the management of one-lung ventilation. Curr Opin Anaesthesiol. 2006 Feb;19(1):1-4. doi: 10.1097/01.aco.0000192778.17151.2c. PMID 16547426
- [Background] Schultz MJ, Haitsma JJ, Slutsky AS, Gajic O. What tidal volumes should be used in patients without acute lung injury? Anesthesiology. 2007 Jun;106(6):1226-31. doi: 10.1097/01.anes.0000267607.25011.e8. PMID 17525599
- [Background] Michelet P, D'Journo XB, Roch A, Doddoli C, Marin V, Papazian L, Decamps I, Bregeon F, Thomas P, Auffray JP. Protective ventilation influences systemic inflammation after esophagectomy: a randomized controlled study. Anesthesiology. 2006 Nov;105(5):911-9. doi: 10.1097/00000542-200611000-00011. PMID 17065884